CLINICAL TRIAL: NCT02414061
Title: The Influence of Whey Protein Addition to a Carbohydrate-based Breakfast on Metabolic and Appetite Parameters Following a Second Meal
Brief Title: Metabolic and Appetite Parameters Following Addition of Whey Protein to a Carbohydrate-based Breakfast
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HLS-13-131017
Record Dates: First submitted 2015-04-07; First posted 2015-04-10 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Healthy
Keywords: Postprandial glycemia; metabolic health measures
MeSH Terms: interventions — Whey Proteins; Breakfast

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Breakfast - Carbohydrate + Whey Protein (Experimental): Addition of whey protein isolate (20 g dissolved in flavoured water) to breakfast meal composition
  Interventions: Dietary Supplement: Whey Protein (Arla Foods Ingredients Group); Other: Breakfast meal
- Breakfast - Carbohydrate (Placebo Comparator): Only flavoured water consumed with breakfast meal
  Interventions: Other: Breakfast meal
- No Breakfast (No Intervention): Only water consumed at breakfast time point

INTERVENTIONS:
Dietary Supplement: Whey Protein (Arla Foods Ingredients Group) — 20 g whey protein isolate added to breakfast meal
  Arms: Breakfast - Carbohydrate + Whey Protein
Other: Breakfast meal — Carbohydrate breakfast served as a standard portion (1799 kJ, 93/2/9% energy from carbohydrate/fat/protein)
  Arms: Breakfast - Carbohydrate; Breakfast - Carbohydrate + Whey Protein

SUMMARY:
The purpose of this study is to investigate whether the addition of whey protein to a breakfast high in carbohydrate content will influence acute metabolic and appetite responses, as well as responses to a subsequent lunch meal.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-40 years old (male)
* Recreationally active (>30 minutes of structured exercise, 5 times/week)

Exclusion Criteria:

* Metabolic disease (e.g. Type 2 diabetes, thyroid disorders)
* Taking any prescribed medication
* Regular breakfast skipper
* Food allergies or intolerances
* Eating disorders
* Smoker

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2014-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Postprandial blood glucose responses | 0-360 minutes post breakfast
  Blood glucose concentration determined in whole blood sampled at regular intervals post-breakfast and post-lunch

SECONDARY OUTCOMES:
Acute subjective appetite responses | 0-360 minutes post breakfast
  Subjective appetite ratings determined from Visual Analogue Scales sampled at regular intervals

CONTACTS AND LOCATIONS:
Overall Officials: Emma J Stevenson, PhD, Study Director — Northumbria University
Locations (1):
- Faculty of Health and Life Sciences, Northumbria University, Newcastle upon Tyne, Tyne and Wear, United Kingdom